CLINICAL TRIAL: NCT04460976
Title: Psychoeducation for Adults With Autism and Their Significant Others/Family Members
Acronym: Prisma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prisma
Record Dates: First submitted 2019-04-08; First posted 2020-07-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Treatment Satisfaction; Knowledge Acquisition Disability Nos; Anxiety; Depression; Quality of Life; Relation, Family; Acceptance of Diagnosis; Stigma of Mental Illness; Participation
Keywords: Autism; Psychoeducation; Adults; Significant others; Knowledge acquisition; Stigma
MeSH Terms: conditions — Anxiety Disorders; Depression; Autistic Disorder; Social Stigma | interventions — mesoglycan; Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Masking at baseline of both participant and care-provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experiment group that receives the psychoeducation direct after the baseline measurement.
  Interventions: Behavioral: Psychoeducation for Adults With Autism and Their Significant Others/Family members (Prisma)
- Control group (Other): Standard care / treatment as usual. Comparison group alos receives Prisma psychoeducation after the three-month follow-up time period.
  Interventions: Behavioral: Treatment as usual/standard care

INTERVENTIONS:
Behavioral: Psychoeducation for Adults With Autism and Their Significant Others/Family members (Prisma) — Psychoeducation in groups
  Arms: Experimental group
Behavioral: Treatment as usual/standard care — Standard care at disability/habilitation services.
  Arms: Control group

SUMMARY:
Prisma is a four-session psychoeducational intervention administered in groups for individuals with ASD together with their family members and significant others. The aspiration is to make Prisma into an affordable, accessible and available intervention. This includes taking into account a great age spectrum, differences in comorbidity as well as other varied qualities that characterize this group. Acknowledging this diversity and helping to create opportunity for these individuals is of great importance in order to follow national as well as international legislations of the patient's rights.

The aim of the proposed studies is to evaluate the feasibility and effect of Prisma in adults (18 or over) with ASD and their family members/significant others in an outpatient clinical habilitation context.

DETAILED DESCRIPTION:
Against the background that interest organizations has identified a need for more knowledge about ASD both in adults with ASD and their significant others, a psychoeducational intervention Prisma was created.

Prisma - the psychoeducational intervention The intervention consists of four 2-hour sessions (2 x 45 min lecture plus paus and time for questions). Two clinicians administer each course and follow a power point with detailed instructions. The goal is to increase knowledge and provide the participants with new insights into their diagnosis and that they get concrete tools that will help them handle obstacles in their everyday life. Another important aspect is to learn more about available support and services.

This research project consists of three studies: An open feasibility study , a randomized controlled trail (RCT) including a three month follow-up, a moderation and mediation study including new outcome variables for stigma and participation.

Study 1. The data collection for the open feasibility study was carried out during the fall of 2017. Data remains to be analyzed. n = 186

Study 2. The RCT will include approximately n=80 in the experimental group and equally many wait-list controls. The RCT also include one significant other per patient which gives a total number of 320 in the RCT. Participants are randomized to be in either the experimental group or the wait-list/treatment as usual controls. The experimental groups receive Prisma according to the manual while the wait-list/TAU controls take part in Prisma approximately 4 months later.

Study 3. In order to expand the analyses beyond what is addressed in the RCT (study 2), researchers would like to investigate if increased knowledge of ASD via participation in Prisma will affect self-stigma and/or affiliate stigma. Importantly, stigma will be investigated both in adults with ASD (self-stigma) and in their significant others (affiliate stigma). Yet another expansion of this project that researchers will address in study 3 is the experiences of active participation and engagement during the Prisma program, and possible association between engagement and treatment results for the adults with ASD and their significant others.This study will include 150 adults with ASD and 150 significant others.

ELIGIBILITY:
Inclusion Criteria:

* Adults with autism spectrum disorder
* Should meet DSM-5 criteria for ASD and/or ICD-10 for one of the autism diagnoses under F84.
* Diagnoses are set within the Swedish healthcare system
* The significant other should also be an adult (18 years or older) and could be a parent, sibling, partner, friend or what the participant with ASD thought of as a significant other.

Exclusion Criteria:

* Intellectual disability.
* Insufficient command of the Swedish language/ unable to understand the content.
* Severe psychiatric comorbidity that made participation difficult (e.g. severe depression, severe suicidality, severe anxiety), other circumstances that could make participation hard (e.g. homelessness) and severe difficulties or discomfort participating in groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Study 1: Evaluation of session 1 | Immediately after intervention
  This includes five items scored on a Likert scale ranging from 0 ("not at all") to 4 ("yes, absolutely"), with item one to three concerning the participants opinion of the content and knowledge acquired and item four to five whether it was useful to trade experiences with the other participants.
  Intervention satisfaction was measured with an evaluation questionnaire after each session, a modified version of the Session evaluation form (SEF: Bramham et al., 2009; Hirvikoski et al., 2017). High values are indication of statisfaction:
  * After today's lecture, my knowledge about ASD has increased
  * I will benefit from what we went through on today's lecture
  * The content of today's lecture felt relevant based on my own experiences
  * It was helpful to be able to share my experiences with other participants
  * It was helpful to take part of others experiences and tips on strategies
Study 1: Evaluation after session 2 | Immediately after intervention
  This includes five items scored on a Likert scale ranging from 0 ("not at all") to 4 ("yes, absolutely"), with item one to three concerning the participants opinion of the content and knowledge acquired and item four to five whether it was useful to trade experiences with the other participants.
  Intervention satisfaction was measured with an evaluation questionnaire after each session, a modified version Session evaluation form (SEF: Bramham et al., 2009; Hirvikoski et al., 2017). High values are indication of statisfaction:
  * After today's lecture, my knowledge about ASD has increased
  * I will benefit from what we went through on today's lecture
  * The content of today's lecture felt relevant based on my own experiences
  * It was helpful to be able to share my experiences with other participants
  * It was helpful to take part of others experiences and tips on strategies
Study 1: Evaluation after session 3 | Immediately after intervention
  This includes five items scored on a Likert scale ranging from 0 ("not at all") to 4 ("yes, absolutely"), with item one to three concerning the participants opinion of the content and knowledge acquired and item four to five whether it was useful to trade experiences with the other participants.
  Intervention satisfaction was measured with an evaluation questionnaire after each session, a modified version of the Session evaluation form (SEF: Bramham et al., 2009; Hirvikoski et al., 2017). High values are indication of statisfaction:
  * After today's lecture, my knowledge about ASD has increased
  * I will benefit from what we went through on today's lecture
  * The content of today's lecture felt relevant based on my own experiences
  * It was helpful to be able to share my experiences with other participants
  * It was helpful to take part of others experiences and tips on strategies
Study 1: Evaluation after session 4 | Immediately after intervention
  This includes five items scored on a Likert scale ranging from 0 ("not at all") to 4 ("yes, absolutely"), with item one to three concerning the participants opinion of the content and knowledge acquired and item four to five whether it was useful to trade experiences with the other participants.
  Intervention satisfaction was measured with an evaluation questionnaire after each session, a modified version of the Session evaluation form (SEF: Bramham et al., 2009; Hirvikoski et al., 2017). High values are indication of statisfaction:
  * After today's lecture, my knowledge about ASD has increased
  * I will benefit from what we went through on today's lecture
  * The content of today's lecture felt relevant based on my own experiences
  * It was helpful to be able to share my experiences with other participants
  * It was helpful to take part of others experiences and tips on strategies
Study 1: Number of individuals that completed the intervention | Immediately after intervention
  To have competed the interevention was measured as attending ≥3 out of 4 sessions
Study 1: Adverse events during the intervention | Through completion of the intervention (typically within 4 weeks)
  (reports of inconvenience or hospitalization due to the intervention)
Study 1: Adverse events after the intervention | Immediately after intervention
  (reports of inconvenience or hospitalization due to the intervention)
Study 1: Overall treatment satisfaction measured by The Evaluation Questionnaire | Immediately after intervention
  The participants (both ASD patient and significant other) also filled out an evaluation form after the last session, a modified version of the Evaluation Questionnaire (Hesslinger et al., 2002; Hirvikoski et al., 2011), about their overall appraisal of the intervention. Higher values are indication of satisfaction. 12 items and was distributed at the end of the last session. Five items regarding the content of the intervention as a whole (i.e. all four group sessions) were scored on a Likert scale ranging from 0-4 (0=not at all, 4= yes, absolutely). ("The content of the intervention has clearly been ASC-related", "My knowledge about ASC has increased", "I am more able to cope with my ASC-related problems", "During the sessions I have been able to give my point of views", "I would attend similar intervention again").The participants also rated the course as a whole following the school grading system ''Failed,'' ''Passed,'' ''Passed with distinction,'' and ''Passed with special
Study 1: Open answer questions regarding Treatment satisfaction measured by The Evaluation Questionnaire | Immediately after intervention
  The participants (patient with ASD and signifcant other) filled out an evaluation form after the last session, a modified version of the Evaluation Questionnaire (Hesslinger et al., 2002; Hirvikoski et al., 2011), about their overall appraisal of the intervention. Higher values are indication of satisfaction. 12 items and was distributed at the end of the last session. Beyond the five items mentioned above, the participants could answer four questions with open answers ("How has the intervention been helpful?", "What could be done to improve the intervention?", "Could you have done anything different?", "Is there anything else you would like to comment?")
Study 1: Well-beining before and after the intervention measures by The Evaluation Questionnaire | Immediately after intervention
  The participants filled out an evaluation form after the last session, a modified version of the Evaluation Questionnaire (Hesslinger et al., 2002; Hirvikoski et al., 2011), about their overall appraisal of the intervention. Since it is of great importance to follow-up the participants well-being, the form contained two items where the participants rated their well-being before and after the intervention ("How would you rate your well-being prior to the intervention?", "How would you rate your current well-being") at T1 and T2 on a scale 1-10 (1= very poor, 10= very good). They could also rate the intervention as whole; answering if they considered it to be "Not approved", "Approved", "Well Approved" or "Very well Approved".
Study 1: Credibility measured with the Credibility Scale (TCS: Borkovec & Nau, 1972) | Immediately after intervention
  Five items: four items that measure treatment credibility and one outcome expectation. Items scored on a 10-point. Likert scale, with a total score range of 0-50. High values = high credibility.
Study 2: Knowledge about autism measured by Autism specific quiz | Change in knowledge from baseline to immediately after the intervention and at three month follow-up
  ASD knowledge was measured using the ASD 20 Questions, a knowledge quiz with 20 true/false/don't know scored items, reflecting knowledge about ASD, which was modified for this study (Bramham et al. 2009; Hirvikoski et al 2017). Total score range from 0-20. High values = more knowledge
Study 3: Participation measured by Patient Participation in Rehabilitation Questionnaire. | Change in knowledge from baseline to immediately after the intervention.
  Active participation during the intervention will be measured with Patient Participation in Rehabilitation Questionnaire (PPRQ: Lindberg et al., 2013). The scale consists of 23 items that are rated on 5 step likert scale. High values = active participation.
Study 3: Patient Stigma | Change from baseline to immediately after the intervention
  Does PRISMA lead to reduced self-stigma for the adult with ASD and/or reduced affiliate stigma for the significant other? The scales we plan to use in study 3 are Internalized Stigma of mental Illness (ISMI) scale (Boyd, Adler, Otilingam & Peters, 2014). The scale consists of 29 items on a 4 step likert scale. High values = more stigma
Study 3: Affiliate Stigma | Change from baseline to immediately after the intervention
  To measure stigma in significant others, we will use Affiliate Stigma scale. This scale is new but show good psychometric properties (Mak & Cheung, 2008). The scale consists of 22 items on a 4 step likert scale. High values = more stigma

SECONDARY OUTCOMES:
All studies: Quality of life: Satisfaction with life scale (SWLS) | Change from baseline to immediately after the intervention and at three month follow-up
  Quality of life is measured with Satisfaction with life scale (SWLS) Pavot & Diener, 1993.
  Its five items are scored on a scale from 1 to 7, indicating very dissatisfied to very satisfied, with 4 as a neutral point.
All studies: Acceptance of diagnosis measured with "What I think about my diagnosis" | Change from baseline to immediately after the intervention and at three month follow-up
  What I think about my diagnosis" for patients with ASD and "What I think about my significant other diagnosis" for significant others. Both questionnaires with 7 items scored on a 7-point likert-scale raging from 1 to 7, "Always true" to "Never true" (Hirvikoski et al, 2017) and based on Acceptance and Action Questionnaire - II (Hayes et al, 2001).
All studies: Well-being with Hospital Anxiety and Depression Scale (HADS) | Change from baseline to immediately after the intervention and at three month follow-up
  The Hospital Anxiety and Depression Scale (A. S. Zigmond & Snaith, 1983) was used to measure well-being on the two subscales Depression and Anxiety containing seven items each, and scored on a 0-3 Likert-scale.
Study 1 and 2: The burden of care on significant others measured with Assessment Scale (BAS) | Change from baseline to immediately after the intervention and at three month follow-up
  The burden of care on significant others was assessed using the Burden Assessment Scale (BAS) (Reinhard et al. 1994), a scale consisting of 19 items scored on a 4-point Likert scale from 1 ("Not at all") to 4 ("A lot").
Study 1 and 2: Relation to significant others (QAFM) | Change from baseline to immediately after the intervention and at three month follow-up
  The Questions About Family Members (QAFM) (Hansson and Jarbin 1997) constitute a dyadic self-report questionnaire, which was used to measure aspects of the quality of the relationship between the co-participants, i.e., the relationship between the adult individual with ASD and his/her significant other(s). The QAFM comprises four subscales: (1) Critical Remarks (directed at the other person); (2) (the respondent's) Emotional Over-involvement; (3) Perceived Criticism (from the other person); and (4) (perceived) Emotional Involvement (from the other person in the relationship). The 30 items are scored on a 1 ("almost never") to 5 ("almost always") Likert scale. Low scores on the first three subscales are indicative of a good quality of relationship, while on the last subscale (Emotional Involvement), high scores indicate the same.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden